CLINICAL TRIAL: NCT05649020
Title: ED50 of Intrathecal Hyperbaric 2% Prilocaine in Transperineal Magnetic Resonance Imaging-Transrectal Ultrasound Fusion Guided Biopsy
Brief Title: ED50 of Intratecal Prilocaine in Ultrasound Fusion Prostate Biopsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Matilde Zaballos, Professor, Hospital General Universitario Gregorio Marañon
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: PRILODE50-FUSION
Record Dates: First submitted 2022-11-30; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Evaluate Requirements of 2% Prilocaine in MR-UF Prostate Biopsy
Keywords: ED50; hyperbaric prilocaine; ultrasound fusion guided prostate biopsy

STUDY DESIGN:
Intervention Model Description: To evaluate the ED50 and ED90 of intrathecal HP for patients undergoing undergoing ambulatory MRI/ultrasound fusión prostate biopsy.
Masking Description: The nurse blinded to the dose, was absent during the procedure and assessed each block. Furthermore, all patients were unaware of the injected dose of HP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prilocaine dose (Other): to determine the ED50 and ED90 of intrathecal HP for patients undergoing undergoing ambulatory MRI/ultrasound fusión prostate biopsy.
  Interventions: Drug: Dose of prilocaine

INTERVENTIONS:
Drug: Dose of prilocaine — With the patient in the sitting position, spinal anesthesia was performed using the midline approach at the L3-L4; L4-L5 interspace with a spinal needle. The dose of HP that a patient received was determined by the previous patient's response. If successful anesthesia was obtained, the next patient's dose was decreased. The first patient will receive a dose of 20 mg. The dose decrement/increment for each subsequent patient will be set at 2 mg. A nurse blinded to the dose, will assess the sensitive level achieved with each block. Furthermore, all patients will be unaware of the injected dose of HP. For purposes of the study, anesthesia was considered successful when there was complete loss of pinprick and cold sensation at the L1 dermatome. Values of ED 50 will be determined by calculating the midpoint concentration after at least 8 crossover points sufficient/insufficient anesthesia will be obtained. A single measurement will be obtained from each patient.
  Other Names: ED50 of intrathecal hyperbaric prilocaine in ultrasound fusion guided prostate biopsy

SUMMARY:
The aim of the present study was to determine the ED50 and ED90 of intrathecal hyperbaric 2% prilocaine (HP) for patients undergoing ambulatory prostate biopsy via magnetic resonance imaging (MRI)/ultrasound fusion.

DETAILED DESCRIPTION:
Prostate biopsy to diagnose or exclude cancer is currently performed an estimated one million times annually worldwide. In this method, the operator images the prostate using ultrasound, as performed for the past several decades; while thus viewing the prostate, the MRI of that prostate, which is performed beforehand and stored in the device, is fused with real-time ultrasound using a digital overlay, allowing the target(s), previously delineated by a radiologist, to be brought into the aiming mechanism of the ultrasound machine. The fusion results in creation of a three-dimensional reconstruction of the prostate, and on the reconstructed model, the aiming and tracking of biopsy sites occurs. This method needs for sedation/general/ spinal anesthesia because of patient discomfort with the transperineal approach of the biopsy needle passing through the perineum.

Even though the MRI/ultrasound fusión prostate biopsy is widespread used, the anaesthetic techniques for this procedure are not standardised. Hyperbaric prilocaine is an amide-type local anesthetic widely used in short surgical procedures showing its efficacy for outpatient surgery. The proposed intrathecal doses of prilocaine for various surgical procedures range from 10 to 80 mg. Thus, even though the drug is in clinical use, optimal doses of HP required for specific types of surgery warrant further refinement. The aim of the present study was to determine the ED50 and ED90 of intrathecal HP for patients undergoing undergoing ambulatory MRI/ultrasound fusión prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

ASA II-III patients Aged 18-85 years Prostate fusion biopsy procedure Scheduled to ambulatory surgery Signed informed consent

Exclusion Criteria:

* Standard contraindications to neuraxial blockade, coagulopathy, site infection, neurological impairment, known allergy to local anesthetics. Refusal of the patient to participate in the study.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
ED50 of intrathecal hyperbaric 2% prilocaine in transperineal magnetic resonance imaging-transrectal ultrasound fusion guided biopsy | From the baseline, previous to prilocaine adminstration until the end of the prostate biopsy procedure. 30 minutes
  to determine the ED50 and ED90 of intrathecal HP for patients undergoing undergoing ambulatory MRI/ultrasound fusión prostate biopsy.

SECONDARY OUTCOMES:
To analyze the hemodynamic response during surgery | From the baseline previous to prilocaine adminstration until the end of the prostate biopsy. 30 minutes
  To evaluate the incidence of hypertension, hypotension, bradycardia or tachycardia during the prostate biopsy procedure.
acute urinary retention | From the baseline previous to prilocaine adminstration until the first 24 hours after the prostate biopsy procedure
  Evaluate the incidence of urinary retention
length of stay in the facility | From the baseline previous to prilocaine adminstration until the patient meets discharge criteria, defined by complete regression of sensory block.
  Time to eligibility for home discharge,
incidence of unplanned admissions | From the baseline previous to prilocaine adminstration until the first 24 hours after the prostate biopsy procedure
  To know the incidence of patients who cannot be discharged from the unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Gregorio Maranon, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan is intended

REFERENCES:
- [Background] Dixon WJ. Staircase bioassay: the up-and-down method. Neurosci Biobehav Rev. 1991 Spring;15(1):47-50. doi: 10.1016/s0149-7634(05)80090-9. PMID 2052197
- [Background] Gebhardt V, Herold A, Weiss C, Samakas A, Schmittner MD. Dosage finding for low-dose spinal anaesthesia using hyperbaric prilocaine in patients undergoing perianal outpatient surgery. Acta Anaesthesiol Scand. 2013 Feb;57(2):249-56. doi: 10.1111/aas.12031. Epub 2012 Nov 30. PMID 23199005
- [Result] Guntz E, Latrech B, Tsiberidis C, Gouwy J, Kapessidou Y. ED50 and ED90 of intrathecal hyperbaric 2% prilocaine in ambulatory knee arthroscopy. Can J Anaesth. 2014 Sep;61(9):801-7. doi: 10.1007/s12630-014-0189-7. Epub 2014 Jun 7. PMID 24906303
- [Result] Camponovo C, Fanelli A, Ghisi D, Cristina D, Fanelli G. A prospective, double-blinded, randomized, clinical trial comparing the efficacy of 40 mg and 60 mg hyperbaric 2% prilocaine versus 60 mg plain 2% prilocaine for intrathecal anesthesia in ambulatory surgery. Anesth Analg. 2010 Aug;111(2):568-72. doi: 10.1213/ANE.0b013e3181e30bb8. Epub 2010 Jun 7. PMID 20529983
- [Result] Boublik J, Gupta R, Bhar S, Atchabahian A. Prilocaine spinal anesthesia for ambulatory surgery: A review of the available studies. Anaesth Crit Care Pain Med. 2016 Dec;35(6):417-421. doi: 10.1016/j.accpm.2016.03.005. Epub 2016 Jun 21. PMID 27352633
- [Result] Forster JG. Short-acting spinal anesthesia in the ambulatory setting. Curr Opin Anaesthesiol. 2014 Dec;27(6):597-604. doi: 10.1097/ACO.0000000000000126. PMID 25211156
- [Result] Hendriks MP, de Weert CJ, Snoeck MM, Hu HP, Pluim MA, Gielen MJ. Plain articaine or prilocaine for spinal anaesthesia in day-case knee arthroscopy: a double-blind randomized trial. Br J Anaesth. 2009 Feb;102(2):259-63. doi: 10.1093/bja/aen357. Epub 2008 Dec 25. PMID 19112061